CLINICAL TRIAL: NCT06416787
Title: A Double Blind, Randomized Study Assessing the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Multiple Ascending Doses of IBI355 in Healthy Volunteers
Brief Title: Safety and Tolerability of IBI355 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CIBI355A103
Record Dates: First submitted 2024-05-11; First posted 2024-05-16 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- IBI355 dose-3 (Experimental): IBI355 15mg/kg and placebo will be given to the subjects every 4 weeks (6:2)
  Interventions: Drug: placebo; Drug: IBI355
- IBI355 dose-1 (Experimental): IBI355 1mg/kg and placebo will be given to the subjects every 4 weeks (6:2)
  Interventions: Drug: placebo; Drug: IBI355
- IBI355 dose-4 (Experimental): IBI355 30mg/kg and placebo will be given to the subjects every 4 weeks (6:2)
  Interventions: Drug: placebo; Drug: IBI355
- IBI355 dose-2 (Experimental): IBI355 7.5mg/kg and placebo will be given to the subjects every 4 weeks (6:2)
  Interventions: Drug: placebo; Drug: IBI355

INTERVENTIONS:
Drug: placebo — IBI355 7.5mg/kg Q4W
Drug: IBI355 — IBI355 1mg/kg Q4W

SUMMARY:
This study aims to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of multiple ascending doses of IBI355 in Healthy volunteers. This study also aims to evaluate the anti-Drug antibody after multiple ascending doses of IBI355 in Healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Understanding and Signing a written informed consent prior to selection;
2. Aged above 18 years old, male or female;
3. Body mass index (BMI) between 18-28kg/m2;
4. Normal label test;
5. No parenting plan for at least 6 months

Exclusion Criteria:

1. Subjects with a history of allergy；
2. Subjects participated in the other clinical trail in 1 month or less than 5 t1/2 since the previous clinical trial (which is longer)；
3. Subjects with an infection requiring systemic medication was present within 30 days prior to randomization;
4. HIV-Ab、RPR、HCV-Ab、HBV、HBeAg or HBcAb, one of them positive;
5. There have a clinical or imaging evidence that the subject with active tuberculosis, or there is evidence that the subject is in the incubation period for tuberculosis;
6. Patients with a history of central nervous system, cardiovascular system, digestive system, respiratory system, urinary system, blood system, metabolic disorders and other systemic diseases;
7. Subject with a hcg positive;
8. Patients with a history of neuropsychiatry or who are considered unfit to participate in this clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2024-05-20 (Actual); Primary Completion 2025-02-26 (Actual); Study Completion 2025-04-02 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events and serious adverse events | Up to week 24

SECONDARY OUTCOMES:
Area under the Curve(AUC) of multi-dose of IBI355 | Up to week 12
Peak serum concentration(Cmax) of multi-dose of IBI355 | Up to week 12
Clearance (CL) of multi-dose of IBI355 | Up to week 12
Half-life (t1/2) of multi-dose of IBI355 | Up to week 12
The ratio of Anti-drug antibody of multi-dose of IBI355 | Up to week 24

CONTACTS AND LOCATIONS:
Locations (1):
- Aerospace Center Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No